CLINICAL TRIAL: NCT00466596
Title: Effect of House Dust Mite Allergen Challenge in Persons Using 1200 mg Gamma Tocopherol Supplements
Acronym: MiteE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Michelle Hernandez, MD, Investigator, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0768
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinitis; Mild Asthma
Keywords: allergic rhinitis; mild asthma; dust mite allergy; gamma tocopherol
MeSH Terms: conditions — Rhinitis, Allergic; Dust Mite Allergy | interventions — gamma-Tocopherol; Vitamin E; Tocopherols; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gamma Tocopherol — 14 days of daily high dose (1200mg) Gamma Tocopherol. Subjects will receive a 14 day supply (28 softgel capsules, approximately 600 grams of gT each) dispensed by the University of North Carolina Hospitals Investigational Drug Service and provided by YASOO Medical.
  Other Names: gT; Vitamin E; Tocopherol; Vitamin

SUMMARY:
Twenty, house dust mite (HDM)-allergic non-smoking subjects with or without mild asthma between the ages 18-50 will be recruited. The primary endpoint will be nasal eosinophilia. Each volunteer will be screened with skin testing, pulmonary function testing and induced sputum. If eligible they will return for baseline nasal allergen challenge and lavage. Approximately two weeks later they will return for gamma tocopherol (gT) dosing visit. After completing 14 days of daily high dose (1200mg) gT, they will return for a second nasal allergen challenge. This visit will also include pulmonary function testing and blood draw. The purpose of this study is to determine if high dose gamma tocopherol therapy can reduce allergen induced nasal inflammation.

DETAILED DESCRIPTION:
This will be done using a single-group, prospective, descriptive proof of concept study design (Phase I) in which HDM-allergic adults will undergo baseline nasal allergen challenge and nasal lavage, then receive 2 weeks of treatment with gT followed by a second challenge and nasal lavage.

Primary outcome: Post-treatment change in concentration of house dust mite-induced eosinophils in nasal lavage fluid (NLF), compared to pre-treatment baseline.

Secondary outcomes: (a) NLF inflammatory mediators including eicosanoid products of COX-2 pathway, inflammatory cytokines relevant to innate immunity and allergic inflammation, cells other than eosinophils including neutrophils, total protein; (b) similar endpoints in induced sputum; (c) sub-analysis of all data for subjects with mild asthma.

Safety outcomes: Post-treatment change in coagulation markers (PT, PTT).

Study Protocol:

Visit 1(Screening): Study subjects consenting for the protocol will be scheduled for an initial baseline screening visit which will include urine pregnancy test, medical history and physical exam, immediate-hypersensitivity skin testing for D. farinae and other common allergens, baseline spirometry, nasal lavage for cell differentials and cytokines, induced sputum for cell differentials and cytokines, venipuncture for up to 30ml of blood for complete blood, count coagulation factors, cytokines and vitamin levels.

Visit 2: Allergen challenge visit will occur within 2 months of screening. Medical history including medications will be reviewed. Urine pregnancy test, physical exam, baseline nasal symptom score will be obtained prior to challenge. Study volunteer will undergo graded nasal allergen challenge with D. farinae using left naris with symptom score recorded after each dose. Nasal allergen challenge will be provided in a graded dose fashion 0 AU, 100 AU, 500 AU and then 1,000 AU separated by 15 minutes. Dilutions will be provided by the University of North Carolina Hospitals Investigational Drug Service. Over 10 minutes, symptoms will be monitored and scored, based on symptoms in the allergen challenge nostril. If there are no positive clinical symptoms, increasing concentrations of dust mite allergen dilution are deposited into the nose. Nasal challenge with saline will be given in the contralateral nostril with similar volumes as used for allergen challenge followed by spirometry and vital signs. Subjects will remain in the research lab and undergo vital signs and spirometry 4 hours post challenge and at the investigator's discretion. Nasal lavage will occur 4 hours after allergen challenge for measurements as noted above. If volunteer was a sputum producer in the first visit, sputum induction will be performed, also 4 hours after nasal allergen challenge. Venipuncture for complete blood count coagulation factors, cytokines and vitamin levels will also be collected.

Visit 2a: This visit will occur within 24 hr after Visit 2. Volunteer will have vital signs recorded, review of symptoms, physical examination and spirometry.

Visit 3(Initial dosing visit): This visit will occur at least 2 weeks after Visit 2. Any changes in medical history, medications or adverse events (AE's) since prior visit will be reviewed. Urine pregnancy test will be performed for females of child bearing potential. Subjects will receive a 14 day supply (28 softgel capsules, approximately 600 grams of gT each) dispensed by the University of North Carolina Hospitals Investigational Drug Service and provided by YASOO Medical. Subjects will be observed while taking the initial oral dose of 2 softgel capsules (approximately 1200 grams) of gT and will be discharged home with individual oral doses of study drug for the following 13 days. Subjects will be given a daily medication diary to record when the dose was taken and any changes in health or medications.

Visit 4: This visit is a safety visit after 6-8 days of gT therapy. The subjects will undergo vital signs measurements, spirometry and physical exam specifically focused on signs of bruising or bleeding. Venipuncture (approximately 10ml) will be performed to obtain CBC and coagulation factors since high dose gT theoretically may affect platelet function and coagulation.

Visit 5: After two weeks of daily gT the subject volunteer will return for another nasal allergen challenge. Medical history will be updated, any AE's or new medications since visit 4 will be reviewed. Pregnancy testing, spirometry and vital signs will be performed. After baseline nasal symptom score is obtained a graded nasal allergen challenge will be performed as in visit 2. Spirometry will be performed after challenge to assure volunteer has tolerated allergen challenge. Nasal lavage will be performed 4 hours after allergen challenge for measurements as noted above. If a volunteer was a sputum producer in previous visit, sputum induction 4 hours after allergen challenge for measurements as above. Venipuncture for blood studies (including safety labs) as indicated in visit above will be performed.

Visit 5a: This visit will occur within 24 hours of Visit 2. Volunteer will undergo vital signs measurement, review of symptoms, physical exam and spirometry.

Visit 6: Five to ten days after challenge, volunteer will return for discontinuation visit which will include vital signs, physical exam and spirometry.

ELIGIBILITY:
Inclusion Criteria:

1. Specific allergy to house dust mite Dermatophagoides farinae confirmed by positive immediate skin test response.
2. Subjects may be enrolled with mild asthma if an FEV1 of at least 80% of predicted and
3. FEV1/FVC ratio of at least .70 (without use of bronchodilating medications for 12 hours), consistent with lung function of persons with mild episodic or mild persistent asthma is demonstrated. For the purpose of this protocol, an asthmatic individual will be defined as having a) positive methacholine challenge with a provocative concentration of methacholine producing a 20% fall in FEV1 (PC20 methacholine) with less than or equal to 10 mg/ml by the method used (see below); OR b) physician diagnosed asthma with symptoms and chronic daily therapy consistent with the mild asthma
4. Ability to withhold antihistamine medications for one week prior to study and one week prior to each nasal challenge visit.
5. Subjects must be able and willing to give informed consent. -

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the allergen challenge study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, bleeding disorder, or chronic thyroid disease.
2. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
3. Use of systemic steroid therapy within the preceding 12 months for treatment of an asthma exacerbation.
4. Use of inhaled or nasal steroids, cromolyn or leukotriene inhibitors (Montelukast or Zafirkulast) within the past month (except for use of cromolyn exclusively prior to exercise).
5. Use of allergen immunotherapy.
6. Use of daily theophylline within the past month.
7. Use of nasal medications that might alter the response to nasal allergen challenge including anti-inflammatory and anti-histamine agents within one week of challenge.
8. Inability to withhold inhaled or oral bronchodilating medications for 12 hours prior to allergen challenge.
9. Pregnancy or nursing a baby.
10. Women of child-bearing age who are not using dependable contraception (such as birth control pills, IUD or estrogen patches) or who are not completely abstinent.
11. Cigarette smoking within the past 12 months of more than 1 pack/week.
12. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
13. Exacerbation of asthma more than 2x/week which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
14. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
15. Viral upper respiratory tract infection within 2 weeks of challenge.
16. Any acute infection requiring antibiotics within 2 weeks of challenge.
17. Participating in an allergen inhalation study within 2 weeks of this challenge or use of any investigational agent within last 30 days.
18. Use of tricyclics or beta-blockers.
19. Use of MAO inhibitors or any medications known to interfere with the treatment of anaphylaxis.
20. Subjects with a history of immunologic disease or undergoing immune suppression for cancer or other diseases.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Post-treatment change in concentration of house dust mite-induced eosinophils in nasal lavage fluid (NLF), compared to pre-treatment baseline. | 4 hours

SECONDARY OUTCOMES:
(a)NLF inflammatory mediators including eicosanoid products, inflammatory cytokines relevant to innate immunity and allergic inflammation, cells other than eosinophils, total protein (b)safety outcomes of cbc and coagulation factors | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Michellle Hernandez, MD, Principal Investigator — University of North Carolina; David B Peden, MS/MD, Study Director — Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Center for Environmental Medicine, Asthma and Lung Biology — http://www.med.unc.edu/cemalb